CLINICAL TRIAL: NCT06055543
Title: Impact of a New Plant-based High-energy Oral Nutritional Supplement on Nutritional Outcomes in Malnourished Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danone Specialized Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fortimel PlantBased Spain 2022
Record Dates: First submitted 2023-09-14; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Malnutrition; Cancer; Inflammatory Bowel Diseases; Chronic Obstructive Pulmonary Disease (COPD); Hiv
MeSH Terms: conditions — Malnutrition; Neoplasms; Inflammatory Bowel Diseases; Pulmonary Disease, Chronic Obstructive; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortimel Energy (Active Comparator): Control: high-energy ONS 1.5 Kcal/m 200ml for 90 days
  Interventions: Dietary Supplement: Fortimel
- Fortimel PlantBased (Experimental): Intervention: high-energy ONS 1.5 Kcal/m 200ml for 90 days
  Interventions: Dietary Supplement: Fortimel

INTERVENTIONS:
Dietary Supplement: Fortimel — 2 bottles/day of the high energy ONS

SUMMARY:
This study aims to compare nutritional outcomes in terms of percentage of weight gain between a new planted-based high-energy ONS and a standard high-energy ONS with animal protein (cow's mil protein) in patients at malnutrition according to Global Leadership Initiative on Malnutrition (GLIM) criteria.

DETAILED DESCRIPTION:
Due to the increasingly pressing need to develop an oral nutritional supplement (ONS) that does not contain animal ingredients, Fortimel PlantBased, suitable for patients with Disease-Related Malnutrition or who wish to avoid or reduce the consumption of animal products for dietary or lifestyle reasons, is being promoted. At the same time, it is also a therapeutic option to be considered in the population with allergy or intolerance to cow's milk protein. Therefore, the aim is to offer an adapted therapeutic nutritional solution that guarantees nutritional results that are not inferior than ONS with animal protein (cow's milk protein).

This study was designed as an open-label randomized controlled non-inferiority trial with two arms: a new planted-based ONS (Fortimel PlantBased) as the intervention arm and standard ONS (Fortimel Energy) as the control arm, both high-energy formulas (1.5 kcal/m; 200ml).

The study will be carried out in patients at malnutrition according to Global Leadership Initiative on Malnutrition (GLIM) criteria, who need to supplement their diet by taking a high-energy ONS for at least 12 weeks. These patients will be treated and follow-up by the Endocrinology and Nutrition services of 6 public hospitals in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old

  * Malnourished patients according to GLIM criteria
  * Patients with a high energy requirement (1.5kcal/ml) requiring the intake of 2 bottles of ONS per day for at least 12 weeks
  * Patients presenting any of the following clinical situations:
* Elderly patients requiring oral nutritional support
* Patients with digestive pathology including but not restricted to inflammatory bowel disease, short bowel syndrome, pancreatitis, without active malabsorption and maldigestion.
* Chronic diseases such as COPD, mild to moderate renal disease, HIV
* Oncologic patients with Eastern Cooperative Oncology Group (ECOG) 0-1

  * Patients who have given their consent to participate
  * Patients who, in the opinion of the physician, have the capacity to answer the study questionnaires themselves or their caregivers

Exclusion Criteria:

* Patients who need ONS due to surgical or acute illness*

  * Patients with known intolerance or allergy to cow's milk, soya or peas
  * Patients with hyperthyroidism. Patients with uncontrolled hypothyroidism
  * Uncontrolled diabetic patients (HbA1c >8%)
  * Patients requiring enteral nutrition by tube or ostomy
  * Patients with moderate and serious renal insufficiency < 30ml/min/1,73 m2
  * Patients who have value creatinine:

    * 1,70 mg/dl - 150,31umol/L Men
    * 1,50 mg/dl - 132,63umol/L Women
  * Patients with levels of haemoglobin <10 g/dl, transferrin <150 mg /dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Changes between baseline and final visit (12 weeks).
  Change in weight percentage
Improvement in nutritional status | From the baseline to the final visit (12 weeks)
  Improvement in nutritional status according to the GLIM criteria. A change in classification category from grade 2 of malnutrition to grade 1 or not meet GLIM criteria, as well as a change from grade 1 to not meet GLIM criteria are considered an improvement.

SECONDARY OUTCOMES:
Change in muscle strength | From the baseline to final visit (12 weeks)
  Measured by dynamometry
Change in calf circumference | From baseline to final visit (12 week)
Percentage of compliance | During the study follow up
  Taking into account the number of bottles per day taken, the ml of product and the ml left over.
Changes in the gastrointestinal symptom scale (GSRS) | From the baseline to final visit (12 week)
  Total score
ONS Satisfaction | Final visit (12 week)
  Patients satisfaction taking ONS will be considered if a patient indicates a score of at least 8 points for overall satisfaction question.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario de Móstoles, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iglesias Hernandez NC, Ramos Carrasco A, De Luis Roman DA, de Pablos-Velasco PL, Calanas Continente A, Rodriguez Soto MJ, Lopez-Gomez JJ, Comi-Diaz C, Garcia-Rey S, Perez-Rambla C, Garcia-Luna PP. Effect of a new plant-based high-energy oral nutritional supplement in adult malnourished patients: an open-label, randomized clinical trial. Front Nutr. 2025 Nov 20;12:1667954. doi: 10.3389/fnut.2025.1667954. eCollection 2025. PMID 41356829